CLINICAL TRIAL: NCT01637506
Title: Correlation Between Excretion Metabolites in Urine and Bacterial Microflora in Patients With Urinary Stone Disease
Brief Title: Urine and Stool Analysis in Kidney Stone Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Ben Chew, MD, Associate Professor, University of British Columbia
Other Study IDs: H10-01195
Record Dates: First submitted 2011-12-13; First posted 2012-07-11 (Estimated); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Urolithiasis
Keywords: urine; stool; kidney stones
MeSH Terms: conditions — Urolithiasis; Kidney Calculi

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — De-identified and study coded urine and stool are collected, processed and analysed in the research laboratory.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Study group: * Age > 19
  * Radiological evidence indicating presence of a current renal or ureteric stone
- Control group: * Age > 19.
  * No history of kidney stone disease

SUMMARY:
The purpose of this study is to add to the investigators' quest to understanding stone disease, by evaluating the metabolites excretion in urine and its relation to microflora present in the stool.

DETAILED DESCRIPTION:
Kidney stones affect up to 10% of the Canadian population and can lead to pain, hospitalization, lost of time at work, and surgery. Approximately 80% of stones consist of calcium and oxalate, of which both components come from diet and normal bodily processes. Individuals who have high levels of oxalate in their urine have a greater tendency to generate stones. One recommendation is to reduce their intake of oxalate-containing foods, but many healthy foods contain oxalate, and an oxalate-free diet is unpalatable and difficult to achieve. Some patients, despite reducing their oxalate intake, still have high amounts in the urine.

Intestinal metabolism is largely affected by the state and composition of the intestinal bacterial flora, with several metabolic diseases being linked to a disrupted "normal" intestinal flora. The investigators believe that calcium oxalate stone disease as well as high urinary levels of oxalate (hyperoxaluria) are triggered by inefficient oxalate metabolism in the intestine, which is linked to a "disrupted" intestinal bacterial flora that lacks certain key components such as O. formigenes. The long-term purpose of this study is therefore, to determine the effect of replenishing the intestinal flora of patients with that of "normal" controls, thereby re-introducing a balanced environment that will lead to the re-establishment of normal metabolic functions and a decrease in urinary oxalate levels and hopefully lower incidence of stone disease.

ELIGIBILITY:
Inclusion Criteria:

Controls

* Age > 19.
* No history of kidney stone disease

Study Patient (Stone Patient)

* Age > 19
* Radiological evidence indicating presence of a current renal or ureteric stone

Exclusion Criteria:

* Pregnancy
* Positive Urine Culture
* Active cancer
* Recurrent urinary infections
* Gross hematuria
* Inability to provide informed consent
* In the Investigator's opinion, the patient would not be good for the study.

Controls Only:

* Family history of kidney stones
* History of kidney stones

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects in the study group are seen at Vancouver General Hospital for their kidney stone disease. Subjects in the control group do not have history or family history of kidney stones and can join the study if they are eligible, wiling to participate, and can provide their specimens at Vancouver General Hospital.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2012-07; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Bacterial flora in the intestine of patients with kidney stones compared to non-stone forming individuals | one day of urine and stool collection
  The objective of this study is to compare the bacterial flora in the intestine of patients with kidney stones compared to non-stone forming individuals. If there are differences between stone forming and non-stone forming individuals in the content of their bacterial flora, these will also be correlated with levels of metabolites found in the urine that are known risk factors of stone disease. Difference in bacterial intestinal flora already exists for patients who are obese compared to non-obese individuals.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Lange, MSc, PhD, Study Director — University of British Columbia; Ryan F Paterson, MD, FRCS(C), Study Director — University of British Columbia; Colin Collins, MA, CA, PhD, Study Director — Vancouver Coastal Health; Stephane LeBihan, PhD, Study Director — Vancouver Prostate Centre
Locations (2):
- Canada (2):
  - Vancouver General Hospital, Vancouver, British Columbia
  - Stone Centre, Vancouver General Hospital, Jim Pattison Pavilion, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No